CLINICAL TRIAL: NCT03712644
Title: Intentional Coronary Revascularization Versus Conservative Therapy in Patients Undergoing Peripheral Artery Revascularization Due to Critical Limb Ischemia
Brief Title: Coronary Revascularization Versus Conservative Therapy in Patients With Treated Critical Limb Ischemia
Acronym: INCORPORATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Gabor Toth-Gayor, Staff-member interventional cardiologist, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30-194 ex 17/18
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Coronary Artery Disease
Keywords: Critical limb ischemia; Coronary artery disease; Fractional flow reserve-guided coronary revascularization
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: non-blinded, open-label, prospective 1:1 randomized controlled multicentric trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative (No Intervention): Patients will receive primarily optimal medical therapy alone and followed, according to protocol. Any further cardiologic investigation will be performed only in case of clinical suspicion of myocardial ischemia related symptoms.
- Invasive (Experimental): In the Invasive group in addition to optimal medical therapy elective coronary angiography will be performed. Coronary catheterization is preferably scheduled within a maximum of 14 days after peripheral revascularization
  All lesions of 50-90% diameter stenosis in a major coronary artery will be evaluated by fractional flow reserve (FFR) and intervened by percutaneous coronary intervention (PCI) if FFR≤0.80 or left for medical therapy if FFR>0.80. All lesions of ≥90% diameter stenosis in a major coronary artery will be intervened. This includes also efforts to recanalize chronic total occlusions (CTO) of large supplied viable myocardial territory.
  For complex cases revascularization by coronary artery bypass surgery might be considered, however PCI is preferred whenever possible.
  Interventions: Device: FFR-guided coronary revascularization

INTERVENTIONS:
Device: FFR-guided coronary revascularization — Stenoses in range of 50-90% diameter stenosis in major coronary arteries will be assessed by FFR, and revascularized if FFR equal to or lower than 0.80. Lesions above 90% diameter stenosis in will be revascularized without further assessment.
  Arms: Invasive

SUMMARY:
The objective of the INCORPORATE trial is to evaluate whether an intentional invasive strategy with ischemia targeted, reasonably complete coronary revascularization and optimal medical therapy is superior as compared to a primary conservative approach and optimal medical therapy alone in terms of spontaneous myocardial infarct-free and overall survival in patients with severe peripheral artery disease, underwent peripheral artery revascularization due to critical limb ischemia.

The INCORPORATE trial is designed to be non-blinded, open-label, prospective 1:1 randomized controlled multicentric trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients, undergoing successful peripheral revascularization (percutaneous or surgical) due to critical limb ischemia will be screened, and enrolled if informed consent form is signed and none of the following exclusion criteria is met.

Exclusion Criteria:

* contraindication for double antiplatelet therapy for at least one month;
* contraindication for guideline-conform longterm antiplatelet/anticoagulation regime after PCI;
* heart failure with ejection fraction below 35%;
* significant valvular heart disease with indication for surgical or percutaneous repair;
* any concomitant disease with a life expectancy less than 2 years;
* severe renal dysfunction with glomerular filtration rate below 30 mL/min/1.73m2;
* ongoing sepsis.

Patients, who cannot be enrolled for any reasons will enter a prospective registry.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of composite of overall death and spontaneous myocardial infarction | 1-year

SECONDARY OUTCOMES:
Rate of composite of overall death and spontaneous myocardial infarction | 2-years
Rate of overall death | 1- and 2-years
Rate of spontaneous myocardial infarction | 1- and 2-years
Quality of life (EQ5D) development | 1- and 2-years
Rate of composite of death, spontaneous myocardial infarction, target coronary revascularization and any stroke | 1- and 2-years
Rate of composite of death, spontaneous myocardial infarction, target coronary revascularization | 1- and 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Gabor G Toth, MD, PhD, Principal Investigator — Div. Cardiology, Dept. Medicine, Medical University Graz, Graz, Austria; Zoltan Ruzsa, MD, PhD, Principal Investigator — Bacs-Kiskun County Hospital, Kecskemet, Hungary; Marianne Brodmann, MD, PhD, Principal Investigator — Div. Angiology, Dept. Medicine, Medical University Graz, Graz, Austria
Locations (2):
- Div. Cardiology and Div. Angiology, Dept. Medicine, Medical University Graz, Graz, Austria
- Bacs-Kiskun County Hospital, Kecskemét, Hungary

REFERENCES:
- [Derived] Toth GG, Brodmann M, Kanoun Schnur SS, Bartus S, Vrsalovic M, Krestianinov O, Kala P, Bil J, Gil R, Kanovsky J, Di Serafino L, Paolucci L, Barbato E, Mangiacapra F, Ruzsa Z. Intentional coronary revascularization versus conservative therapy in patients after peripheral artery revascularization due to critical limb ischemia: the INCORPORATE trial. Clin Res Cardiol. 2025 Aug;114(8):991-999. doi: 10.1007/s00392-024-02487-2. Epub 2024 Jul 11. PMID 38990250
- [Derived] Toth G, Brodmann M, Barbato E, Mangiacapra F, Schneller L, Orias V, Gil R, Bil J, Bartus S, Ruzsa Z. Rational and design of the INtentional COronary revascularization versus conservative therapy in patients undergOing successful peripheRAl arTEry revascularization due to critical limb ischemia trial (INCORPORATE trial). Am Heart J. 2019 Aug;214:107-112. doi: 10.1016/j.ahj.2019.05.005. Epub 2019 May 16. PMID 31200280